CLINICAL TRIAL: NCT02178696
Title: Predictors of Antidepressant Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jon-Kar Zubieta, MD PhD, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HUM00033328
Record Dates: First submitted 2014-06-12; First posted 2014-07-01 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Citalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Known Placebo First (Experimental): This arm gets a placebo that they know is a placebo (called inactive), then has 2 scans performed (FMRI and PET), then a 2-3 day washout, and then gets a so-called "active medication" (which is also actually a placebo), and another pair of scans. Following these, participants receive 10 weeks of open-label antidepressant administration (Celexa or alternative as explained in intervention description). First line antidepressant will be Celexa unless not clinically indicated.
  Interventions: Other: Placebo, identified as placebo to participants; Drug: Celexa or other antidepressant as clinically indicated; Other: Placebo, identifed to participants as "Active medication"
- "Active" (blinded) Placebo first group (Experimental): This arm gets a placebo that they don't know is a placebo (called Active), then has 2 scans performed (FMRI and PET), then a 2-3 day washout, and then gets a so-called "inactive medication" (which participants know is a placebo), and another pair of scans. Following these, participants receive 10 weeks of open-label antidepressant administration (Celexa as explained in intervention description). First line antidepressant will be Celexa unless not clinically indicated.
  Interventions: Other: Placebo, identified as placebo to participants; Drug: Celexa or other antidepressant as clinically indicated; Other: Placebo, identifed to participants as "Active medication"

INTERVENTIONS:
Other: Placebo, identified as placebo to participants — White tablets
Drug: Celexa or other antidepressant as clinically indicated — Open label s-citalopram, 20 mg start up dose, increasing to 40 mg as clinically indicated; If prior non-response to this medication is noted by the patient, alternative treatments may include another first-line antidepressant:fluoxetine 20 mg; paroxetine up to 60 mg; sertraline up to 200 mg; bupropion up to 300 mg
  Other Names: S-citalopram 20-40 mg orally
Other: Placebo, identifed to participants as "Active medication" — Blue Capsule

SUMMARY:
Major depression is a highly prevalent, frequently debilitating illness that too often fails to respond to currently available treatments such as antidepressant medication. Furthermore, randomized controlled trials of antidepressants consistently demonstrate large placebo effects. The investigators hypothesize that individual differences in the function of key brain circuits underlie the observed variability in clinical responses to both placebo and antidepressant medication. This study will test this hypothesis by recruiting treatment-seeking volunteers with major depression, with or without comorbid nicotine dependence. Volunteers will participate in positron emission tomography (PET) and functional magnetic resonance imaging (fMRI) scans in the context of a treatment trial in which they will receive both placebo and antidepressant medication. A major goal of the study is to improve prediction of individual clinical responses in future treatment trials in which brain imaging may be unavailable, and to study the mechanisms of antidepressant response in Major Depression.

DETAILED DESCRIPTION:
We performed a single-blinded two-week cross-over randomized controlled trial of two identical oral placebos (described as having either potentially "active" fast-acting antidepressant-like effects or to be "inactive") followed by a 10-week open-label treatment with a selective serotonin reuptake inhibitor (SSRI) or in some cases, another agent as clinically indicated. The volunteers were studied with PET and the µ-opioid receptor selective radiotracer [11C]carfentanil after each 1-week "inactive" and "active" oral placebo treatment. In addition, 1 mL of isotonic saline was administered intravenously (i.v.) within sight of the volunteer during PET scanning every 4 min over 20 min only after the 1-week active placebo treatment, with instructions that the compound may be associated with the activation of brain systems involved in mood improvement. This challenge stimulus was utilized to test the individual capacity to acutely activate endogenous opioid neurotransmission under expectations of antidepressant effect.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria will include:

* Participants diagnosed with Major Depressive Disorder and will include Hamilton Depressive Rating Scale (HDRS) scores >15

Exclusion Criteria:

* Comorbid conditions that are medical, neurological or psychiatric, pregnancy, use of hormones (including birth control) or use of psychotropic agents
* We will only permit certain past anxiety disorder diagnoses, including generalized anxiety, panic, agoraphobia, social phobia
* We also will exclude left-handed individuals and patients who have used any centrally acting medications or recreational drugs with the past 2 months
* No history of an implant, pacemaker or pacemaker wires, open heart surgery, artificial heart valve, brain aneurysm surgery, middle ear implant, hearing aid, braces or extensive dental work, cataract surgery or lens implant, implanted mechanical or electrical device, or artificial limb or joint
* No metallic object in their body (such as braces) or have a history of foreign metallic object in the body such as bullets, BB's, pellets, shrapnel, or other metal fragments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon-Kar Zubieta, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- Department of Psychiatry, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Pecina M, Bohnert AS, Sikora M, Avery ET, Langenecker SA, Mickey BJ, Zubieta JK. Association Between Placebo-Activated Neural Systems and Antidepressant Responses: Neurochemistry of Placebo Effects in Major Depression. JAMA Psychiatry. 2015 Nov;72(11):1087-94. doi: 10.1001/jamapsychiatry.2015.1335. PMID 26421634
- [Result] Sikora M, Heffernan J, Avery ET, Mickey BJ, Zubieta JK, Pecina M. Salience Network Functional Connectivity Predicts Placebo Effects in Major Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2016 Jan;1(1):68-76. doi: 10.1016/j.bpsc.2015.10.002. PMID 26709390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 consented volunteers dropped because of exclusion criteria
Pre-assignment Details: Of 44 participants consented, 4 were not assigned to participate due to screen failures.
Period: First Assignment and Washout
Arm/Group | Known Placebo First | "Active" (Blinded) Placebo First Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Assignment After Crossover
Arm/Group | Known Placebo First | "Active" (Blinded) Placebo First Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Open-label Antidepressant
Arm/Group | Known Placebo First | "Active" (Blinded) Placebo First Group
Started | 20 | 20
Completed | 14 | 13
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Population: Because this is a crossover study, the entire population is represented together for baseline measures
Arm/Group | Total Study Population
Number analyzed (Participants) | 40
Age, Customized [Count of Participants; unit: Participants]
  19 to 59 years | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Changes in Mu-opioid Binding Potential During PET
Description: Binding Potential = Bmax/Kd (receptor concentration/affinity). This is the most common measure of in vivo receptor binding with positron emission tomography. Whole brain changes in mu-opioid receptors binding potential during PET from the Inactive to the Active placebo condition.
  Positive numbers presented here represent reductions in binding potential from the inactive to the active condition.
Time Frame: (90 minute PET scans) assessed at Weeks 1 and 2
Population: Data in four subjects was missing due to failure in the synthesis of the radio tracer for at least one of the two scans.
Measure: Mean (Standard Deviation); unit: Binding potential ratio
Groups:
- Changes in Mu-opioid Binding (Inactive -Active Placebo): Average regional changes in mu-opioid binding potential from the Inactive to the Active Placebo Condition.
Arm/Group | Changes in Mu-opioid Binding (Inactive -Active Placebo)
Number analyzed (Participants) | 36
Binding potential ratio | 0.12 (0.32)
Statistical Analysis 1: Comparison: Changes in Mu-opioid Binding (Inactive -Active Placebo); Test type: Other; p < 0.001, t-test, 2 sided — A p<0.001 was established for regions a priori hypothesized (e.g. nucleus accumbens); Mean Difference (Net) = 0.12, 95% CI 2-sided [0.016 to 0.23], Standard Deviation 0.31

2. Primary Outcome: Changes in BOLD Response During Reward fMRI Task (Monetary Incentive Delay, MID)
Description: % BOLD signal changes in the nucleus accumbens from the Inactive to the Active Placebo condition.
Time Frame: (90 minute fMRI scans) assessed at Weeks 1 and 2
Population: Data was missing in 11 subjects due to movement artifacts, or incidental findings that made the data not usable.
Measure: Mean (Standard Deviation); unit: % BOLD changes from Inactive to Active
Groups:
- Changes in BOLD Responses During the MID After Placebo: Changes in BOLD response from the Inactive to the Active condition during the Monetary Incentive Delayed Task in the Nucleus Accumbens.
Arm/Group | Changes in BOLD Responses During the MID After Placebo
Number analyzed (Participants) | 29
% BOLD changes from Inactive to Active | 0.04 (1.13)

3. Secondary Outcome: Changes in Dopamine (D 2/3) Binding Potential During PET.
Description: Binding Potential= Bmax/Kd (receptor concentration/affinity). This is the most common measure of in vivo receptor binding with PET.
  Striatal changes in D2/3 receptor binding potential during PET from the Inactive to the Active condition.
  Positive numbers presented here represented reductions in binding potential from the inactive to the active condition.
Time Frame: (90 minute PET scan) assessed at Weeks 1 and 2
Population: Data was only collected in 26 subjects as proposed.
Measure: Mean (Standard Deviation); unit: Binding potential ratio
Groups:
- Average Regional Changes in D2/3 Binding (Inactive-Active Plac: Average regional changes in D2/3 binding potential from the Inactive to the Active placebo condition.
Arm/Group | Average Regional Changes in D2/3 Binding (Inactive-Active Plac
Number analyzed (Participants) | 26
Binding potential ratio | 0.08 (0.15)

4. Secondary Outcome: Changes From Baseline in Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16) Score
Description: This scale is a self-report measure of depression with 16 items.
  Questions in the QIDS - SR-116 correlate with the nine DSM-IV symptom criterion domains, Including: Sleep disturbance (initial, middle, and late insomnia or hypersomnia) (Q 1 - 4), Sad mood (Q 5), Decrease/increase in appetite/weight (Q 6 - 9), Concentration (Q 10), Self-criticism (Q 11), Suicidal ideation (Q 12), Interest (Q 13), Energy/fatigue (Q 14), Psychomotor agitation/retardation (Q 15 - 16).
  Severity of depression can be judged based on the total score: 1-5= No depression; 6-10= Mild depression; 11-15= Moderate depression; 16-20= Severe depression; 21-27= Very severe depression.
  The PHQ-9 and QIDS were used to assess changes in mood during the placebo intervention (first 2 weeks), and therefore results are described as changes from the inactive to the active condition.
Time Frame: From Pre to post- active placebo, and from pre to post- inactive placebo (1 week intervention)
Population: Changes in QIDS-16SR from screening active/inactive placebo condition to the post scan active/inactive placebo condition.
  Approximately 1-2 weeks between the two conditions.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Active Placebo | Inactive Placebo
Number analyzed (Participants) | 40 | 40
Units on a scale | 1.7 (3.3) | -0.5 (3.2)

5. Secondary Outcome: Changes From Baseline in PHQ-9 Depression Scores.
Description: The Patient Health Questionnaire-9, is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression, based on participant answers. PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression, respectively. The minimum possible score is 0 and the maximum possible score is 27.
  The PHQ-9 and QIDS were used to assess changes in mood during the placebo intervention (first 2 weeks), and therefore results are described as changes from the inactive to the active condition.
Time Frame: From Pre to post- active placebo, and from pre to post- inactive placebo (1 week intervention)
Population: Changes in PHQ-9 score from the beginning of the active/inactive placebo and the end of active/inactive PET scan.
  Approximately 1-2 weeks between the two conditions.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Active Placebo | Inactive Placebo
Number analyzed (Participants) | 40 | 40
Units on a scale | 1.6 (3.6) | 0.96 (3.9)

6. Secondary Outcome: Hamilton Depression Rating Scale Scores
Description: The total score is obtained by summing the score of each item, 0-4 (symptom is absent, mild, moderate, or severe) or 0-2 (absent, slight or trivial, clearly present). For the 17-item version, scores can range from 0 to 54, with 0 meaning no depression, and 54, severe depression.
  The Hamilton Depression Rating Scale was used to assess symptoms during the open label antidepressant treatment phase, so results are described as mean scores at each bi-weekly visit.
Time Frame: Screening, week 0, week 2, week 4, week 8 and week 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Antidepressant Treatment After Placebo Experiment
Number analyzed (Participants) | 40
Units on a scale
  Screening | 21 (4.4)
  week 0 | 17.2 (6.5)
  week 2 | 13.3 (7.18)
  Week 4 | 11 (7.73)
  week 8 | 8.65 (6.78)
  week 10 | 5.3 (3.75)

7. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Designed in 1979 by researchers as an adjunct to the Hamilton Rating Scale for Depression (HAMD) which would be more sensitive to the changes brought on by antidepressants and other forms of treatment than the Hamilton Scale. MADRS was used to assess symptoms during the open label antidepressant treatment phase, so results are described as mean scores at each bi-weekly visit.
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60 where 0 is no depression and 60 is most extreme depression.
  The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
  Usual cutoff points are:
  0 to 6 - normal[5] /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Time Frame: Screening, week 0, week 2, week 4, week 8 and week 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MADRS Scores During the Open-label Antidepressant Treatment
Number analyzed (Participants) | 40
Units on a scale
  Baseline | 27 (6.6)
  week 0 | 22 (8.4)
  week 2 | 15 (7)
  week 4 | 13 (10)
  week 8 | 11 (9.7)
  week 10 | 7.7 (5.36)

ADVERSE EVENTS:
Time Frame: 13 weeks per person
Arm/Group | Placebo (Unknown) | Known Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes